CLINICAL TRIAL: NCT00238654
Title: A Multicenter, Open-Label, Two-Arm Prospective Study to Evaluate the Impact of Patient Readiness to Self-Inject on Outcomes When Using the Copaxone® Prefilled Syringes [The "READY" Trial]
Brief Title: A Study to Evaluate Readiness to Self-inject on Adherence and Compliance to Copaxone® Therapy
Status: Completed | Type: Observational
Sponsor: Teva Neuroscience, Inc. (Industry)
Responsible Party: Thomas Smith, M.D., Vice President, Medical Affairs, Teva Neuroscience
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Other Study IDs: PM08
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study has patients responding to two sets of surveys that will tell their doctor or nurse about their readiness to begin self-injection. In addition, patients will have their self-injection observed and evaluated on up to three visits

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years of age or older, with diagnosis of RRMS
2. Naive to treatment or previously treated with an IFN.

Exclusion Criteria:

1. Not eligible for treatment based on clinical criteria and current indication.
2. Unable to respond to surveys or provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RRMS patient with treatment-naïve or treatment-experienced
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2003-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Adherence of self-injection assessed by self-report at each follow-up visit | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: MerriKay Oleen-Burkey, Ph.D., Study Director — Teva Neuroscience, Inc.